CLINICAL TRIAL: NCT07171021
Title: The Effect of Oral Theophylline on Traumatic Anosmia: A Prospective, Randomized Clinical Trial
Brief Title: The Effect of Oral Theophylline on Traumatic Anosmia
Acronym: theophylline
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Taichung Veterans General Hospital (Other)
Responsible Party: Principal Investigator, Rong-San Jiang, Visiting Doctor, Taichung Veterans General Hospital
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: CF20317A; TCVGH-1117310C (Other Grant/Funding Number: Taichung Veterans General Hospital)
Record Dates: First submitted 2025-09-05; First posted 2025-09-12 (Actual); Last update posted 2025-09-12 (Actual); Status verified 2025-09

CONDITIONS: Traumatic Anosmia
Keywords: olfactory training, smell identification, smell threshold, theophylline, traumatic anosmia
MeSH Terms: interventions — Theophylline; Olfactory Training

STUDY DESIGN:
Who Masked: Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- theophylline arm (Experimental): theophylline (400 mg twice a day) and olfactory training for 6 months
  Interventions: Drug: Theophylline 200 mg; Behavioral: olfactory training
- control arm (Active Comparator): olfactory training for 6 months
  Interventions: Behavioral: olfactory training

INTERVENTIONS:
Drug: Theophylline 200 mg — taking theophylline (400 mg twice a day) and performing olfactory training for 6 months
  Arms: theophylline arm
Behavioral: olfactory training — performing olfactory training for 6 months

SUMMARY:
This study aimed to improve the treatment outcomes of patients with post-traumatic anosmia through medication and olfactory training. Number of subjects and selection criteria: 160 patients were enrolled in the ENT and head and neck outpatient clinic with a history of head trauma, a complaint of anosmia, and evidence of olfactory examination. Their olfactory status had not improved after steroids, zinc tablets, and olfactory training. Exclusion criteria: Patients under 20 years of age, pregnant or breastfeeding women, and those with compromised immune systems were excluded.

Patients who did not improve after medication and olfactory training were randomized. One group received theophylline and zinc tablets with continued olfactory training, while the other group received zinc tablets alone with continued olfactory training. Patients returned for follow-up and medical consultation after treatment at the 24th week. Theophylline medication: Theophylline (200 mg, two tablets twice daily) was administered for 24 weeks.

DETAILED DESCRIPTION:
We collected subjects who complained of a complete loss of their smell function (anosmia) after an episode of head injury between December 2020 and December 2023. Any patient who had a history of loss of olfactory function before head trauma or sinus surgery was excluded from the study. If the etiology of loss of olfactory function was suspected to not be caused by head trauma, it was also excluded. The remaining patients received right and left unilateral phenyl ethyl alcohol (PEA) odor detection threshold tests to assess their olfactory function. The definition of anosmia in this study was that the unilateral PEA thresholds for the right and left were -1. Anosmic patients were included in this study. These anosmic patients were then treated with high-dose prednisolone (1 mg/kg per day for 3 days) with tapering, along with zinc gluconate (10 mg three times a day) for a period of 1 month. Classic OT using 4 separate bottles of PEA, lemon, eucalyptus, and clove oil was also started. The patients were told to sniff each odorant for 10 seconds, twice a day.21 After one month of treatment, all patients received unilateral right and left PEA odor detection threshold tests and the traditional Chinese version of the University of Pennsylvania Identification Test (UPSIT-TC) to assess their olfactory function. Those whose unilateral PEA thresholds on the right and left remained -1 were enrolled in this study.

The eligible patients were randomly divided into 2 groups. Randomized assignment to the two groups was performed by an independent statistician. The patients in the theophylline group took theophylline (400 mg twice a day) for 6 months and continued OT. Those who were assigned to the OT group continued OT for 6 months without any other form of treatment.

All patients returned to the clinic to receive another series of unilateral right and left PEA threshold tests and UPSIT-TC at the end of 6 months of treatment. Patients taking oral theophylline also received blood tests to measure blood theophylline levels. Brain magnetic resonance imaging (MRI) was performed to measure the volumes of olfactory bulbs (OB) following completion of the 6-month treatment. During the 6-month treatment period, drugs such as oral or nasal steroids, vitamin A, zinc, and antihistamines were not allowed.

ELIGIBILITY:
Inclusion Criteria:

* subjects who complained of a complete loss of their smell function (anosmia) after an episode of head injury.

Exclusion Criteria:

* patients without a complete loss of their smell function
* a history of loss of olfactory function before head trauma or sinus surgery
* the etiology of loss of olfactory function was suspected to not be caused by head trauma

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 158 (Actual)
Dates: Start 2020-12-01 (Actual); Primary Completion 2023-12-31 (Actual); Study Completion 2024-06-30 (Actual)

PRIMARY OUTCOMES:
Change of olfactory identification ability of participants with treatment as assessed by Traditional Chinese Version of the University of Pennsylvania Identification Test | From enrollment to the end of treatment at 7 months
  The test consists of 40 tests as it follows the North American version of the University of Pennsylvania Smell Identification Test. In each test, the brown strip at the bottom of the test page consists of microcapsules of an odorant that are released by scratching the strip with a pencil tip. The patient sniffs the released odorant and selects a response from four odor descriptor options that are used to identify the odorant. The test score is the number of correct responses among the 40 tests taken.
Olfactory threshold change of participants with intervention drug as assessed by phenyl ethyl alcohol odor detection threshold test | From enrollment to the end of the treatment at 7 months
  The test uses different concentrations of a phenyl ethyl alcohol odorant to measure a patient's odor detection threshold. The strongest concentration is a concentration of phenyl ethyl alcohol at 10-1 log vol/vol. Then, the concentration of the odorant is diluted with mineral oil in half-log steps until the weakest concentration at 10-9 log vol/vol. A 2-alternative forced choice single-staircase procedure is used to decide the odor detection threshold. The threshold ranges from -1 to -9.

CONTACTS AND LOCATIONS:
Locations (1):
- Taichung Veterans General Hospital, Taichung, Taiwan

IPD SHARING:
Plan to Share IPD: Yes
all IPD that underlie results in a publication
Supporting Information: Study Protocol, SAP, ICF
Time Frame: October 2025- October 2025
Access Criteria: Request to Central contact person

REFERENCES:
- [Background] Henkin RI, Velicu I, Schmidt L. An open-label controlled trial of theophylline for treatment of patients with hyposmia. Am J Med Sci. 2009 Jun;337(6):396-406. doi: 10.1097/MAJ.0b013e3181914a97. PMID 19359985